CLINICAL TRIAL: NCT03612076
Title: Cost of Failure Following Reimplantation After a 2-stage Exchange Strategy for Hip or Knee Prosthetic Joint Infection
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Heraeus Medical GmbH (Unknown)
Responsible Party: Sponsor
Other Study IDs: 17-089
Record Dates: First submitted 2018-07-27; First posted 2018-08-02 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Prosthetic Joint Infection
Keywords: prosthetic joint infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Global cost of management of PJI
  Interventions: Other: Global cost of management of PJI

INTERVENTIONS:
Other: Global cost of management of PJI — estimation of the global cost to manage PJI with 2-step exchange over 3 years

SUMMARY:
This study concerns patients having had an infection on their prosthesis (hip, knee,..) and for whom a 2-step exchange of prosthesis has been done.

A 2-step exchange consists in explantation of the prosthesis and implementation of a spacer at the first stage, and reimplantation of a new prosthesis in a second stage. Patients with late prosthetic joint infection are at risk for superinfection at the time of reimplantation.

The aim of this study is to determine the global cost of management of prosthetic joint infection.

ELIGIBILITY:
Inclusion Criteria:

* patients with prosthetic joint infection having had a 2-step exchange and managed at the CRIOAc from at least the reimplantation (between 2013 and 2015)

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with prosthetic joint infection having had a 2-step exchange.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Global cost of management of PJI | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption)
  The following data are collected : duration of hospitalization at the Croix Rousse hospital (surgery unit, department of infectiology, other…) and in post-acute care structures, bacteriology, surgeries, medical treatments… and all acts realized throughout the management of the PJI.

CONTACTS AND LOCATIONS:
Overall Officials: Tristan Ferry, Md,PhD, Principal Investigator — Hospices Civils de Lyon - Hôpital de la Croix-Rousse
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided